CLINICAL TRIAL: NCT02928653
Title: The Effect of Low Calorie Sweetener Consumption on Body Weight, Body Composition, Appetite, and Energy Intake
Brief Title: Beverage Consumption and Fine Motor Control
Acronym: LCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor of Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 055-044
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Body Weight
Keywords: energy intake; energy expenditure; appetite
MeSH Terms: conditions — Body Weight | interventions — Beverages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sucrose Sweetened Beverage (Active Comparator): 100-140 g sucrose/day
  Interventions: Dietary Supplement: Beverage
- Aspartame Sweetened Beverage (Experimental): 0.541-0.757 g aspartame Sweetened Beverage/day
  Interventions: Dietary Supplement: Beverage
- Saccharin Sweetened Beverage (Experimental): 0.300-0.455 g saccharin Sweetened Beverage/day
  Interventions: Dietary Supplement: Beverage
- Sucralose Sweetened Beverage (Experimental): 0.167-0.233 g sucralose Sweetened Beverage/day
  Interventions: Dietary Supplement: Beverage
- Rebaudioside A Sweeteened Beverage (Experimental): 0.250-0.350 g rebaudioside A Sweetened Beverage/day
  Interventions: Dietary Supplement: Beverage

INTERVENTIONS:
Dietary Supplement: Beverage — Participants will receive 1.25 - 1.75 L of sweetened beverage a day for 12 weeks

SUMMARY:
The aim of this study will be to compare the effects of daily consumption of aspartame, rebaudioside a, saccharin, sucralose, and sucrose on body weight and composition in a standardized protocol. The investigators hypothesize that individual low calorie sweeteners (consumed in a beverage) differ from each other in promoting weight loss and decreased fat mass (without energy restriction or dietary guidance) based on their chemical structure.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-40 kg/M2
* Non or rare users of LCS
* Willing to consume large volumes of beverages daily

Exclusion Criteria:

* Weight change > 3kg in the last year
* Plan to initiate a new diet plan in the next 6 months
* Exhibit eating restraint
* Pregnant/lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2015-12; Primary Completion 2018-02 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks
Body Composition | 12 weeks
  Duel emission X-ray absorbtiometry
Energy Intake | 12 weeks
  24 hr Dietary Recall
Appetite | 12 weeks
  24 hr visual analog scale appetite
Energy Expenditure | 12 weeks
  accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Higgins KA, Mattes RD. A randomized controlled trial contrasting the effects of 4 low-calorie sweeteners and sucrose on body weight in adults with overweight or obesity. Am J Clin Nutr. 2019 May 1;109(5):1288-1301. doi: 10.1093/ajcn/nqy381. PMID 30997499